CLINICAL TRIAL: NCT01643746
Title: C-arm CT Evaluation of Luminal Expansion in Stenting Severe Femoro-popliteal Atherosclerotic Disease: Supera Versus LifeStent
Brief Title: Evaluation of Luminal Expansion Following Stenting of Femoro-popliteal Occlusive Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study has never started. The sponsor has decided to not move forward
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Abbott Medical Devices (Industry); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 12.048
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Femoropopliteal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Supera stent (Active Comparator): The Supera stent is a novel interwoven nitinol stent design with high flexibility and radial strength. The radial force of the Supera stent is 4 times higher than comparable nitinol stent.
  Interventions: Device: Supera Stent
- LifeStent (Active Comparator): LifeStent is likely the best reference nitinol stent for comparison because a low restenosis rate has been reported at 1 year with low target revascularization.
  Interventions: Device: Life Stent

INTERVENTIONS:
Device: Supera Stent — Angioplasty and stenting will performed according to the guidelines of the Society of Interventional Radiology and the instruction for use for each stent. Patients will be allocated to Supera stent versus LifeStent based on block randomization (block size 4 patients).
  Arms: Supera stent
Device: Life Stent — Angioplasty and stenting will performed according to the guidelines of the Society of Interventional Radiology and the instruction for use for each stent. Patients will be allocated to Supera stent versus LifeStent based on block randomization (block size 4 patients).
  Arms: LifeStent

SUMMARY:
The primary goal of this trial is to compare prospectively stent opening of Supera (IDEV Technologies) versus a reference stent (LifeStent, Bard Medical) using C-arm CT. A secondary goal is to correlate stent opening with stent patency as documented by Doppler ultrasound at one year post implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient (or legally authorized representative) must give a written informed consent.
* Symptomatic peripheral-artery disease with moderate or severe intermittent claudication and failure of medical treatment (Rutherford stage 2,3) or chronic critical limb ischemia with pain while the patient is at rest (Rutherford stage 4) or chronic critical limb ischemia with ischemic ulcers (Rutherford stage 5, 6) and stenosis of more than 70 percent or occlusion of the ipsilateral superficial femoral artery and/or proximal popliteal artery with a target-lesion length of ≥ 8 and ≤ 20 cm and at least one patent (less than 50 percent stenosed) tibioperoneal runoff vessel (TASC A,B,C lesions)25. Proximal popliteal artery is defined as the popliteal artery above the joint line. The distal portion of the lesion should be located at least 4 cm above the joint line and the distal end of the stent 2 cm above the joint line.
* ABI ≤ 0.9 at rest. Toe-Brachial Index (TBI) may be used if ABI is inadequate.
* Lesion with a calcification percentage of at least 25% based on CTA evaluation (within 6 months of patient enrolment)

Exclusion Criteria:

* Acute critical limb ischemia
* Untreated inflow disease of the ipsilateral pelvic arteries (more than 50 percent stenosis or occlusion).
* Renal failure, creatinine clearance < 50 µmol /l
* Severe allergy to iodine contrast
* Patients with uncorrected bleeding disorders or patients who cannot receive anticoagulation or antiplatelet aggregation therapy
* Lesions < 8 and > 20 cm in length
* Calcification volume of less than 25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Stent expansion | At the completion of the intervention
  Difference in minimal lumen diameter (MLD), minimal lumen area (MLA) and incomplete stent expansion as defined by C-arm CT between both groups

SECONDARY OUTCOMES:
Stent patency | 1 year
  Correlate stent opening with stent patency as documented by Doppler ultrasound at one year post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Soulez, MD, MSc, Study Director — Centre hospitalier de l'université de Montreal
Locations (2):
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Centre hospitalier de l'université de Montréal, Montreal, Quebec